CLINICAL TRIAL: NCT03417492
Title: Cerebrovascular Reactivity Assessed With Functional Near-infrared Spectroscopy and Magnetic Resonance Imaging as a Biomarker of Traumatic Microvascular Injury in American Football Players
Brief Title: Cerebrovascular Reactivity in American Football Players
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty enrolling participants due to COVID emergency, and planned start of new study to address this question in a more rigorous fashion.
Sponsor: University of Pennsylvania (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Presidential Professor, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 827103
Record Dates: First submitted 2017-10-11; First posted 2018-01-31 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Traumatic Brain Injury; Mild Traumatic Brain Injury; Post-Concussion Syndrome
Keywords: TBI; CVR; Hypercapnia; fNIRS; functional magnetic resonance imaging (fMRI); American football
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Post-Concussion Syndrome; Hypercapnia | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Open-label, non-placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sildenafil Citrate (Experimental): Open label treatment with forced titration of sildenafil citrate.
  Interventions: Drug: Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil Citrate — Three 20 mg capsules for the single dose studies. For the 5-week treatment phase, subjects will be assigned to a titration of doses for the 5 week duration of the study. Subjects will be instructed to take 20mg twice per day for 3 days, then 40mg twice per day for 3 days, and then 80mg twice per day for 4 weeks.
  Other Names: Open label forced titration with sildenafil citrate.

SUMMARY:
Investigators will measure cerebrovascular reactivity (CVR) using functional near-infrared spectroscopy (fNIRS) and magnetic resonance imaging (MRI) during the chronic phase after repetitive mild traumatic brain injury (rmTBI) as a biomarker of traumatic cerebrovascular injury (TCVI). We hypothesize that CVR will be decreased in patients with rmTBI and that these decreases will correlate with clinical outcomes. Furthermore, we predict that 5 week administration of a phosphodiesterase 5 (PDE5) inhibitor, sildenafil citrate, will augment CVR in patients with a history rmTBI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-65 years
2. Former National Football League (NFL) players or former varsity college football players
3. Ability to undergo MRI scanning
4. Ability to read, write, and speak English
5. Stable doses of concomitant medications for last 2 weeks prior to enrollment
6. Diagnosis of post-concussive syndrome according to Diagnostic and Statistical Manual 5 (DSM-5) criteria

Exclusion Criteria:

1. Contraindication to sildenafil
2. Past medical history or evidence of penetrating brain injury
3. Daily therapy with a PDE5 inhibitor within the past 2 months, or taken as needed within past 4 weeks
4. History or evidence of pre-existing disabling neurological or psychiatric disorder not related to previous head injuries
5. History of melanoma
6. History of diagnosed obstructive/ restrictive pulmonary disease 7 .) Contraindication to MRI

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Effect of single dose sildenafil citrate treatment on global blood oxygen level-dependent (BOLD) response to hypercapnia. | Immediate
  Determine if single dose treatment with sildenafil (60 mg orally) is effective in increasing the global BOLD response to hypercapnia (5% CO2).

SECONDARY OUTCOMES:
Effect of single dose sildenafil citrate treatment on functional near-infrared spectroscopy (fNIRS) response to hypercapnia. | Immediate
  Determine if single dose treatment with sildenafil (60 mg orally) is effective in increasing the functional near-infrared spectroscopy (fNIRS) response to hypercapnia (5% CO2).
Maximum tolerable dose of sildenafil therapy without severe adverse events. | 5 weeks
  The number of participants reporting treatment-related adverse events (AEs) and serious adverse events (SAEs) will be monitored after each dose increase. AEs and SAEs are assessed using CTCAE, v4.0.

OTHER OUTCOMES:
Effect of 5 weeks sildenafil treatment on CVR as measured by BOLD response to hypercapnia. | 5 weeks
  To evaluate the effects of 5 weeks of treatment on CVR by measuring BOLD signal in response to hypercapnia after 5 week treatment with sildenafil, compared to within-subject CVR response before sildenafil treatment.
Effect of 5 weeks sildenafil treatment on CVR as measured by fNIRS response to hypercapnia. | 5 weeks
  To evaluate the effects of 5 weeks of treatment on CVR by measuring fNIRS signal in response to hypercapnia after 5 week treatment with sildenafil, compared to within-subject CVR response before sildenafil treatment.
Effect of 5 weeks of sildenafil treatment on attention using Trail Making Test Part A. | 5 weeks
  To evaluate the effects of 5 weeks of treatment with sildenafil citrate on attention, measured using the Trail Making Test Part A.
Effect of 5 weeks of sildenafil treatment on attention using the Digit Symbol Modalities Test. | 5 weeks
  To evaluate the effects of 5 weeks of treatment with sildenafil citrate on attention, measured using the Digit Symbol Modalities Test.
Effect of 5 weeks of sildenafil treatment on executive function using the Trail Making Test Part B. | 5 weeks
  To evaluate the effects of 5 weeks of treatment with sildenafil citrate on executive function, measured using the Trail Making Test Part B.
Effect of 5 weeks of sildenafil treatment on executive function using the Neuropsychological Assessment Battery (NAB) mazes. | 5 weeks
  To evaluate the effects of 5 weeks of treatment with sildenafil citrate on executive function, measured using the Neuropsychological Assessment Battery (NAB) mazes.
Effect of 5 weeks of sildenafil treatment on executive function using the Controlled Oral Word Association Test (COWAT). | 5 weeks
  To evaluate the effects of 5 weeks of treatment with sildenafil citrate on executive function, measured using the Controlled Oral Word Association Test (COWAT).
Effect of 5 weeks of sildenafil treatment on language and memory using the Animal Fluency test. | 5 weeks
  To evaluate the effects of 5 weeks of treatment with sildenafil citrate on language and memory, measured using the Animal Fluency test.
Effect of 5 weeks of sildenafil treatment on language and memory using the NAB List Learning test. | 5 weeks
  To evaluate the effects of 5 weeks of treatment with sildenafil citrate on language and memory, measured using the NAB List Learning test.
Effect of 5 weeks of sildenafil treatment on daily function using the Functional Activities Questionnaire. | 5 weeks
  To evaluate the effects of 5 weeks of treatment with sildenafil citrate on daily function, measured using the Functional Activities Questionnaire. The questionnaire requires the subject to rate the level of difficulty/dependency of each task listed (rating range from 0-3). A lower score indicates less difficulty in the listed activities while a higher score indicates more difficulty. The ratings are summed and the total score is reported (range 0-30).

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States